CLINICAL TRIAL: NCT01526265
Title: Way to Quit - Comparative Efficacy, Acceptance and Effectiveness of Health Incentive Structures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Scott Halpern, Assistant Professor of Medicine and Epidemiology , Division of Pulmonary and Critical Care Medicine, Senior Fellow, Center for Bioethics & Leonard Davis Institute of Health Economics, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 814761; R01CA159932 (NIH)
Record Dates: First submitted 2012-01-31; First posted 2012-02-03 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Tobacco Use Disorder
Keywords: Smoking Cessation; Work-site; Incentives; Health Behavior; Smoking
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Health Behavior; Smoking

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Usual Care (Active Comparator): Participants will be offered free smoking cessation programs, and be provided web-based education regarding the health and economic benefits of smoking cessation. Participants will also have the opportunity to submit weekly reports on their smoking habits. They will be informed that they will receive reimbursements for completing the surveys that are part of the Way To Quit program and for submitting saliva or urine samples at 14 days, 30 days, 6 months, and 12 months (among those eligible).
  Interventions: Behavioral: Usual Care
- Individual Rewards (Experimental): Same as USUAL CARE arm, plus financial incentive as follows: if participants quit smoking by their target quit date, and that is confirmed by cotinine or anabasine tests, they will receive a monetary award from the study investigators.
  Interventions: Behavioral: Individual Rewards
- Fixed Deposits (Experimental): Same as USUAL CARE arm, plus financial incentive as follows: participants will have to deposit a certain monetary amount of their own money as an incentive to quit smoking. If they quit smoking by their target quit date, and that is confirmed by cotinine or anabasine tests, participants will receive their deposit back. If participants do not quit, their money will be used to support future research studies designed to help people stop smoking. As a motivation to quit smoking, the participant's deposit will be matched by the study investigators in a rate of 3:1.
  Interventions: Behavioral: Fixed Deposits
- Competitive Deposits (Pari-Mutuel) (Experimental): Same as USUAL CARE, plus financial incentive as follows: groups (or "cohorts") of 6 smokers each will be formed on a rolling basis, linking individuals with target quit dates (day "0's") near each other. Participants will deposit a certain monetary amount (Y) in an account, which will be matched on a rate of 3:1 by the study investigators (M), and the payout for quitting on this arm will be (Y+M) x 6/Q , where Q is the number of quits in the cohort. Again, success will be confirmed by cotinine or anabasine tests, and if participants do not quit, their money will be used to support future research studies designed to help people stop smoking.
  Interventions: Behavioral: Competitive Deposits (Pari-Mutuel)
- Collaborative Rewards (Experimental): Same as USUAL CARE arm, plus financial incentive as follows: groups (or "cohorts") of 6 smokers each will be formed on a rolling basis, linking individuals with target quit dates (day "0's") near each other. If participants quit smoking by their target quit date, and that is confirmed by cotinine or anabasine tests, they will receive a monetary award from the study investigators. On top of that, participants will receive an additional monetary amount for each member of their group who also quits smoking. These participants will interact through a chat room, which will help motivate them to quit smoking.
  Interventions: Behavioral: Collaborative Rewards

INTERVENTIONS:
Behavioral: Usual Care — Participants will receive reimbursements for completing the surveys that are part of the Way To Quit program and for submitting saliva or urine samples at 14 days, 30 days, 6 months, and 12 months (among those eligible).
  Arms: Usual Care
Behavioral: Individual Rewards — If participants quit smoking by their target quit date, and that is confirmed by cotinine/anabasine tests, they will receive a monetary award from the study investigators.
  Arms: Individual Rewards
Behavioral: Fixed Deposits — Participants will have to deposit a certain monetary amount of their own money as an incentive to quit smoking. If they quit smoking by their target quit date, and that is confirmed by cotinine/anabasine tests, participants will receive their deposit back. If participants do not quit, their money will be used to support future research studies designed to help people stop smoking. As a motivation to quit smoking, the participant's deposit will be matched by the study investigators in a rate of 3:1.
  Arms: Fixed Deposits
Behavioral: Competitive Deposits (Pari-Mutuel) — Groups (or "cohorts") of 6 smokers each will be formed on a rolling basis, linking individuals with target quit dates (day "0's") near each other. Participants will deposit a certain monetary amount (Y) in an account, which will be matched on a rate of 3:1 by the study investigators (M), and the payout for quitting on this arm will be (Y+M) x 6/Q , where Q is the number of quits in the cohort. Again, success will be confirmed by cotinine or anabasine tests, and if participants do not quit, their money will be used to support future research studies designed to help people stop smoking.
  Arms: Competitive Deposits (Pari-Mutuel)
Behavioral: Collaborative Rewards — Groups (or "cohorts") of 6 smokers each will be formed on a rolling basis, linking individuals with target quit dates (day "0's") near each other. If participants quit smoking by their target quit date, and that is confirmed by cotinine or anabasine tests, they will receive a monetary award from the study investigators. On top of that, participants will receive an additional monetary amount for each member of their group who also quits smoking. These participants will interact through a chat room, which will help motivate them to quit smoking.
  Arms: Collaborative Rewards

SUMMARY:
Using the NIH-funded Way to Health platform, the investigators will conduct this smoking cessation randomized controlled trial (RCT) among CVS employees. The investigators will be able to determine the comparative and absolute efficacy and effectiveness of 4 different incentive structures that are each grounded in behavioral economic principles. Additionally, the investigators will measure rates of and reasons for acceptance of each incentive structure, and examine participant characteristics that modify the efficacy and acceptance of different incentive structures.

DETAILED DESCRIPTION:
Specific Aim I: Compare the efficacy and effectiveness of 4 financial incentive structures for improving "quit rates" (rates of prolonged smoking abstinence for 6 months): (a) individual financial rewards, (b) individual deposit contracts, (c) cooperative rewards, and (d) competitive deposit contracts

H1: Compared with usual care, all 4 incentive structures will increase quit rates significantly.

H2: Compared with individual financial rewards of equivalent size and schedule, individual deposit contracts, cooperative rewards, and competitive contracts will each increase quit rates significantly.

H3: Group-oriented structures will increase quit rates significantly more than individual-oriented structures.

Specific Aim II: Compare smokers' acceptance of these 4 financial incentive structures for smoking cessation

H4: Uptake rates of reward-based structures will be higher than of structures involving deposit contracts.

H5: Uptake rates of group-oriented structures will be higher than of individual-oriented structures.

Specific Aim III: Identify individual characteristics that modify incentive structures' efficacy and acceptance

H6: Incentives will promote relatively greater quit rates among participants with fewer substitute reinforcers.

H7: Incentives will promote relatively greater quit rates among participants with lower incomes.

H8: Higher-income persons will be relatively more likely to accept incentives requiring deposit contracts.

ELIGIBILITY:
Inclusion Criteria:

* Active smoker of 5 cigarettes per day for at least 6 months;
* At least 18 years old;
* Current full- or part-time employee of CVS or be a family member or friend of a current full- or part-time employee of CVS.

Exclusion Criteria:

* Use a form of tobacco other than cigarettes while participating in the study (as this may influence biochemical testing);
* Are unable or unwilling to access the internet;
* Are unable to provide informed consent.
* Due to the web-based nature of this study, people without reliable computer and internet access will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2185 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Salivary cotinine or anabasine testing (metabolites of nicotine) | at 6 months following the patient selected target quit date.
  The primary measure of smoking cessation will be prolonged abstinence for 6 months, which will be measured by salivary cotinine testing or by urinary anabasine testing (for those participants using nicotine replacement therapy). Saliva samples will be analyzed using semi-quantitative immunochromatographic assay test strips at the University of Pennsylvania. Urine samples will be analyzed using gas chromatography at the Associated Regional and University Pathologists (ARUP) Lab, at the University of Utah.

SECONDARY OUTCOMES:
Salivary cotinine or anabasine testing (metabolites of nicotine) | at 14 and 30 days, and 6 months following the patient selected target quit date and relapse rate 12 months after the target quit date.
  Another secondary outcome variable will be the proportion of participants achieving point prevalence abstinence at 14 days, 30 days, 6 months and 12 months after the quit date.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Halpern, MD, Ph.D., Principal Investigator — University of Pennsylvania, Department of Medicine, Pulmonary, Allergy and Critical Care; Kevin Volpp, MD, Ph.D., Principal Investigator — University of Pennsylvania; Benjamin French, MS, Ph.D., Principal Investigator — University of Pennsylvania; Dylan Small, Ph.D., Principal Investigator — University of Pennsylvania; David Asch, MD, MBA, Principal Investigator — University of Pennsylvania; Janet Audrain-McGovern, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Audrain J, Boyd NR, Roth J, Main D, Caporaso NF, Lerman C. Genetic susceptibility testing in smoking-cessation treatment: one-year outcomes of a randomized trial. Addict Behav. 1997 Nov-Dec;22(6):741-51. doi: 10.1016/s0306-4603(97)00060-9. PMID 9426791
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Background] Pomerleau CS, Carton SM, Lutzke ML, Flessland KA, Pomerleau OF. Reliability of the Fagerstrom Tolerance Questionnaire and the Fagerstrom Test for Nicotine Dependence. Addict Behav. 1994 Jan-Feb;19(1):33-9. doi: 10.1016/0306-4603(94)90049-3. PMID 8197891
- [Background] Hymowitz N, Cummings KM, Hyland A, Lynn WR, Pechacek TF, Hartwell TD. Predictors of smoking cessation in a cohort of adult smokers followed for five years. Tob Control. 1997;6 Suppl 2(Suppl 2):S57-62. doi: 10.1136/tc.6.suppl_2.s57. PMID 9583654
- [Background] Kenford SL, Fiore MC, Jorenby DE, Smith SS, Wetter D, Baker TB. Predicting smoking cessation. Who will quit with and without the nicotine patch. JAMA. 1994 Feb 23;271(8):589-94. doi: 10.1001/jama.271.8.589. PMID 8301790
- [Background] Halpern SD, Madison KM, Volpp KG. Patients as mercenaries?: the ethics of using financial incentives in the war on unhealthy behaviors. Circ Cardiovasc Qual Outcomes. 2009 Sep;2(5):514-6. doi: 10.1161/CIRCOUTCOMES.109.871855. No abstract available. PMID 20031885
- [Background] Giuffrida A, Torgerson DJ. Should we pay the patient? Review of financial incentives to enhance patient compliance. BMJ. 1997 Sep 20;315(7110):703-7. doi: 10.1136/bmj.315.7110.703. PMID 9314754
- [Background] Delmonico FL, Arnold R, Scheper-Hughes N, Siminoff LA, Kahn J, Youngner SJ. Ethical incentives--not payment--for organ donation. N Engl J Med. 2002 Jun 20;346(25):2002-5. doi: 10.1056/NEJMsb013216. No abstract available. PMID 12075064
- [Background] Dickert N, Grady C. What's the price of a research subject? Approaches to payment for research participation. N Engl J Med. 1999 Jul 15;341(3):198-203. doi: 10.1056/NEJM199907153410312. No abstract available. PMID 10403861
- [Background] Macklin R. On paying money to research subjects: 'due' and 'undue' inducements. IRB. 1981 May;3(5):1-6. No abstract available. PMID 11649367
- [Background] Volpp KG, Troxel AB, Pauly MV, Glick HA, Puig A, Asch DA, Galvin R, Zhu J, Wan F, DeGuzman J, Corbett E, Weiner J, Audrain-McGovern J. A randomized, controlled trial of financial incentives for smoking cessation. N Engl J Med. 2009 Feb 12;360(7):699-709. doi: 10.1056/NEJMsa0806819. PMID 19213683
- [Background] Halpern SD, Karlawish JH, Casarett D, Berlin JA, Asch DA. Empirical assessment of whether moderate payments are undue or unjust inducements for participation in clinical trials. Arch Intern Med. 2004 Apr 12;164(7):801-3. doi: 10.1001/archinte.164.7.801. PMID 15078651
- [Background] Halpern SD, Raz A, Kohn R, Rey M, Asch DA, Reese P. Regulated payments for living kidney donation: an empirical assessment of the ethical concerns. Ann Intern Med. 2010 Mar 16;152(6):358-65. doi: 10.7326/0003-4819-152-6-201003160-00005. PMID 20231566
- [Background] DiClemente CC, Prochaska JO, Fairhurst SK, Velicer WF, Velasquez MM, Rossi JS. The process of smoking cessation: an analysis of precontemplation, contemplation, and preparation stages of change. J Consult Clin Psychol. 1991 Apr;59(2):295-304. doi: 10.1037//0022-006x.59.2.295. PMID 2030191
- [Background] Prochaska JO, DiClemente CC, Velicer WF, Rossi JS. Standardized, individualized, interactive, and personalized self-help programs for smoking cessation. Health Psychol. 1993 Sep;12(5):399-405. doi: 10.1037//0278-6133.12.5.399. PMID 8223364
- [Background] Brownson RC, Eriksen MP, Davis RM, Warner KE. Environmental tobacco smoke: health effects and policies to reduce exposure. Annu Rev Public Health. 1997;18:163-85. doi: 10.1146/annurev.publhealth.18.1.163. PMID 9143716
- [Background] Audrain-McGovern J, Rodriguez D, Epstein LH, Rodgers K, Cuevas J, Wileyto EP. Young adult smoking: what factors differentiate ex-smokers, smoking cessation treatment seekers and nontreatment seekers? Addict Behav. 2009 Dec;34(12):1036-41. doi: 10.1016/j.addbeh.2009.06.012. Epub 2009 Jul 5. PMID 19619948
- [Background] Audrain-McGovern J, Rodriguez D, Epstein LH, Cuevas J, Rodgers K, Wileyto EP. Does delay discounting play an etiological role in smoking or is it a consequence of smoking? Drug Alcohol Depend. 2009 Aug 1;103(3):99-106. doi: 10.1016/j.drugalcdep.2008.12.019. Epub 2009 May 14. PMID 19443136
- [Background] Bickel WK, Odum AL, Madden GJ. Impulsivity and cigarette smoking: delay discounting in current, never, and ex-smokers. Psychopharmacology (Berl). 1999 Oct;146(4):447-54. doi: 10.1007/pl00005490. PMID 10550495
- [Background] Johnson MW, Bickel WK, Baker F. Moderate drug use and delay discounting: a comparison of heavy, light, and never smokers. Exp Clin Psychopharmacol. 2007 Apr;15(2):187-94. doi: 10.1037/1064-1297.15.2.187. PMID 17469942
- [Background] Kirby KN, Petry NM, Bickel WK. Heroin addicts have higher discount rates for delayed rewards than non-drug-using controls. J Exp Psychol Gen. 1999 Mar;128(1):78-87. doi: 10.1037//0096-3445.128.1.78. PMID 10100392
- [Background] Baker F, Johnson MW, Bickel WK. Delay discounting in current and never-before cigarette smokers: similarities and differences across commodity, sign, and magnitude. J Abnorm Psychol. 2003 Aug;112(3):382-92. doi: 10.1037/0021-843x.112.3.382. PMID 12943017
- [Background] Pocock SJ, Simon R. Sequential treatment assignment with balancing for prognostic factors in the controlled clinical trial. Biometrics. 1975 Mar;31(1):103-15. PMID 1100130
- [Background] Westman EC, Behm FM, Simel DL, Rose JE. Smoking behavior on the first day of a quit attempt predicts long-term abstinence. Arch Intern Med. 1997 Feb 10;157(3):335-40. PMID 9040302
- [Background] Efron B. International Symposium on Hodgkin's Disease. Session 6. Survival data and prognosis. Invited discussion: Forcing a sequential experiment to be balanced. Natl Cancer Inst Monogr. 1973 May;36:571-2. No abstract available. PMID 4582998
- [Background] Brown CH, Ten Have TR, Jo B, Dagne G, Wyman PA, Muthen B, Gibbons RD. Adaptive designs for randomized trials in public health. Annu Rev Public Health. 2009;30:1-25. doi: 10.1146/annurev.publhealth.031308.100223. PMID 19296774
- [Background] Volpp KG, Pauly MV, Loewenstein G, Bangsberg D. P4P4P: an agenda for research on pay-for-performance for patients. Health Aff (Millwood). 2009 Jan-Feb;28(1):206-14. doi: 10.1377/hlthaff.28.1.206. PMID 19124872
- [Background] Lussier JP, Heil SH, Mongeon JA, Badger GJ, Higgins ST. A meta-analysis of voucher-based reinforcement therapy for substance use disorders. Addiction. 2006 Feb;101(2):192-203. doi: 10.1111/j.1360-0443.2006.01311.x. PMID 16445548
- [Background] Burns DM, Shanks T, Major J, Gower KB, Shopland D. Restrictions on Smoking in the Workplace: Smoking and Tobacco Control Monograph No. 12. Bethesda, MD: National Institutes of Health, U.S. Department of Health and Human Services, National Cancer Institute; 2002.
- [Background] MacPhillamy DJ, Lewinsohn PM. Manual for the pleasant events schedule. Eugene, OR: University of Oregon; 1976.
- [Background] Chapman GB. Time discounting of health outcomes In: Loewenstein G, Read D, Baumeister R, eds. Time and decision: Economic and psychological perspectives on intertemporal choice. New York, NY: Russell Sage Foundation; 2003:395-417.
- [Background] Frederick S, Loewenstein G, O'Donoghue T. Time discounting and time preference: a Critical Review. Journal of Economic Literature 2002;40(2):351-401.
- [Background] True Random Number Service. (Accessed April 6, 2010, at www.random.org.)
- [Background] Dragalin V. Adaptive designs: Terminology and classification. Drug Information Journal 2006;40(4):425-35.
- [Background] Kahneman D, Tversky A. Prospect theory: An analysis of decision under risk. Econometrica 1979;47:263-91.
- [Background] Thaler RH. Some empirical evidence on time inconsistency. Review of Economic Studies 1981;23:165-80.
- [Background] Thaler RH. Mental Accounting and Consumer Choice. Marketing Science 1985;4:199-214.
- [Background] Higgins ST, Heil SH, Dantona R, Donham R, Matthews M, Badger GJ. Effects of varying the monetary value of voucher-based incentives on abstinence achieved during and following treatment among cocaine-dependent outpatients. Addiction. 2007 Feb;102(2):271-81. doi: 10.1111/j.1360-0443.2006.01664.x. PMID 17222282
- [Background] Mokdad AH, Marks JS, Stroup DF, Gerberding JL. Actual causes of death in the United States, 2000. JAMA. 2004 Mar 10;291(10):1238-45. doi: 10.1001/jama.291.10.1238. PMID 15010446
- [Background] Centers for Disease Control and Prevention (CDC). State-specific smoking-attributable mortality and years of potential life lost--United States, 2000-2004. MMWR Morb Mortal Wkly Rep. 2009 Jan 23;58(2):29-33. PMID 19165137
- [Background] Hatsukami DK, Stead LF, Gupta PC. Tobacco addiction. Lancet. 2008 Jun 14;371(9629):2027-38. doi: 10.1016/S0140-6736(08)60871-5. PMID 18555914
- [Background] Centers for Disease Control and Prevention (CDC). Cigarette smoking among adults and trends in smoking cessation - United States, 2008. MMWR Morb Mortal Wkly Rep. 2009 Nov 13;58(44):1227-32. PMID 19910909
- [Background] Hughes JR. Motivating and helping smokers to stop smoking. J Gen Intern Med. 2003 Dec;18(12):1053-7. doi: 10.1111/j.1525-1497.2003.20640.x. PMID 14687265
- [Background] U.S. Department of Health and Human Services. Healthy People 2010: Understanding and Improving Health. Washington, DC: U.S. Department of Health and Human Services; 2000.
- [Background] Hennrikus DJ, Jeffery RW, Lando HA, Murray DM, Brelje K, Davidann B, Baxter JS, Thai D, Vessey J, Liu J. The SUCCESS project: the effect of program format and incentives on participation and cessation in worksite smoking cessation programs. Am J Public Health. 2002 Feb;92(2):274-9. doi: 10.2105/ajph.92.2.274. PMID 11818305
- [Background] Donatelle R, Hudson D, Dobie S, Goodall A, Hunsberger M, Oswald K. Incentives in smoking cessation: status of the field and implications for research and practice with pregnant smokers. Nicotine Tob Res. 2004 Apr;6 Suppl 2:S163-79. doi: 10.1080/14622200410001669196. PMID 15203819
- [Background] Volpp KG, Gurmankin Levy A, Asch DA, Berlin JA, Murphy JJ, Gomez A, Sox H, Zhu J, Lerman C. A randomized controlled trial of financial incentives for smoking cessation. Cancer Epidemiol Biomarkers Prev. 2006 Jan;15(1):12-8. doi: 10.1158/1055-9965.EPI-05-0314. PMID 16434580
- [Background] Coffield AB, Maciosek MV, McGinnis JM, Harris JR, Caldwell MB, Teutsch SM, Atkins D, Richland JH, Haddix A. Priorities among recommended clinical preventive services. Am J Prev Med. 2001 Jul;21(1):1-9. doi: 10.1016/s0749-3797(01)00308-7. PMID 11418251
- [Background] Cromwell J, Bartosch WJ, Fiore MC, Hasselblad V, Baker T. Cost-effectiveness of the clinical practice recommendations in the AHCPR guideline for smoking cessation. Agency for Health Care Policy and Research. JAMA. 1997 Dec 3;278(21):1759-66. PMID 9388153
- [Background] Newhouse JP, McClellan M. Econometrics in outcomes research: the use of instrumental variables. Annu Rev Public Health. 1998;19:17-34. doi: 10.1146/annurev.publhealth.19.1.17. PMID 9611610
- [Background] Angrist A, Imbens G, Rubin D. Identification of Causal Effects Using Instrumental Variables. Journal of the American Statistical Association 1996;91:444-55.
- [Background] Hu FF, Zhang LX, He XM. Efficient Randomized-Adaptive Designs. Annals of Statistics 2009;37(5A):2543-60.
- [Background] Hughes JR, Keely JP, Niaura RS, Ossip-Klein DJ, Richmond RL, Swan GE. Measures of abstinence in clinical trials: issues and recommendations. Nicotine Tob Res. 2003 Feb;5(1):13-25. PMID 12745503
- [Background] Higgins ST, Bickel WK, Hughes JR. Influence of an alternative reinforcer on human cocaine self-administration. Life Sci. 1994;55(3):179-87. doi: 10.1016/0024-3205(94)00878-7. PMID 8007760
- [Background] Silverman K, Chutuape MA, Bigelow GE, Stitzer ML. Voucher-based reinforcement of cocaine abstinence in treatment-resistant methadone patients: effects of reinforcement magnitude. Psychopharmacology (Berl). 1999 Sep;146(2):128-38. doi: 10.1007/s002130051098. PMID 10525747
- [Background] Schotter A, Weigelt K. Behavioral Consequences of Corporate Incentives and Long-Term Bonuses - an Experimental-Study. Manage Sci 1992;38(9):1280-98.
- [Background] Connolly T, Butler DU. Regret in Economic and Psychological Theories of Choice. Journal of Behavioral Decision Making 2006;19(2):148-58.
- [Background] Hoelzl E, Loewenstein G. Wearing out your shoes to prevent someone else from stepping into them: Anticipated regret and social takeover in sequential decisions. Organizational Behavior and Human Decision Processes 2005;98:15-27.
- [Background] Petry NM, Martin B, Cooney JL, Kranzler HR. Give them prizes, and they will come: contingency management for treatment of alcohol dependence. J Consult Clin Psychol. 2000 Apr;68(2):250-7. doi: 10.1037//0022-006x.68.2.250. PMID 10780125
- [Background] Hall SM, Delucchi KL, Velicer WF, Kahler CW, Ranger-Moore J, Hedeker D, Tsoh JY, Niaura R. Statistical analysis of randomized trials in tobacco treatment: longitudinal designs with dichotomous outcome. Nicotine Tob Res. 2001 Aug;3(3):193-202. doi: 10.1080/14622200110050411. PMID 11506764
- [Background] Hosmer DW, Lemeshow S. Model building strategies and methods for logistic regression. In: Hosmer DW, Lemeshow S, eds. Applied Logistic Regression, 2nd Edition. New York: John Wiley & Sons; 2000.
- [Background] Greenland S, Schwartzbaum JA, Finkle WD. Problems due to small samples and sparse data in conditional logistic regression analysis. Am J Epidemiol. 2000 Mar 1;151(5):531-9. doi: 10.1093/oxfordjournals.aje.a010240. PMID 10707923
- [Background] Pagoto SL, Kozak AT, John P, Bodenlos JS, Hedeker D, Spring B, Schneider KL. Intention-to-treat analyses in behavioral medicine randomized clinical trials. Int J Behav Med. 2009;16(4):316-22. doi: 10.1007/s12529-009-9039-3. PMID 19319693
- [Background] Have TR, Joffe MM, Lynch KG, Brown GK, Maisto SA, Beck AT. Causal mediation analyses with rank preserving models. Biometrics. 2007 Sep;63(3):926-34. doi: 10.1111/j.1541-0420.2007.00766.x. PMID 17825022
- [Background] Ten Have TR, Elliott MR, Joffe M, Zanutto E, Datto C. Causal models for randomized physician encouragement trials in treating primary care depression. Journal of the American Statistical Association 2004;99(465):16-25.
- [Background] Small DS, Ten Have TR, Joffe MM, Cheng J. Random effects logistic models for analysing efficacy of a longitudinal randomized treatment with non-adherence. Stat Med. 2006 Jun 30;25(12):1981-2007. doi: 10.1002/sim.2313. PMID 16220487
- [Background] Ten Have TR, Joffe M, Cary M. Causal logistic models for non-compliance under randomized treatment with univariate binary response. Stat Med. 2003 Apr 30;22(8):1255-83. doi: 10.1002/sim.1401. PMID 12687654
- [Background] Guo WS, Ratcliffe SJ, Ten Have TT. A random pattern-mixture model for longitudinal data with dropouts. Journal of the American Statistical Association 2004;99(468):929-37.
- [Background] Giacomini MK, Cook DJ. Users' guides to the medical literature: XXIII. Qualitative research in health care A. Are the results of the study valid? Evidence-Based Medicine Working Group. JAMA. 2000 Jul 19;284(3):357-62. doi: 10.1001/jama.284.3.357. PMID 10891968
- [Background] Strauss AL, Corbin J. Basics of Qualitative Research: Techniques and Procedures for Developing Grounded Theory. Thousand Oaks, CA: Sage; 1998.
- [Background] Charmaz K. Constructing grounded theory: a practical guide through qualitative analysis. Thousand Oaks, CA: Sage Publications; 2006.
- [Background] Bradley EH, Curry LA, Devers KJ. Qualitative data analysis for health services research: developing taxonomy, themes, and theory. Health Serv Res. 2007 Aug;42(4):1758-72. doi: 10.1111/j.1475-6773.2006.00684.x. PMID 17286625
- [Derived] Theodoulou A, Fanshawe TR, Leavens E, Theodoulou E, Wu AD, Heath L, Stewart C, Nollen N, Ahluwalia JS, Butler AR, Hajizadeh A, Thomas J, Lindson N, Hartmann-Boyce J. Differences in the effectiveness of individual-level smoking cessation interventions by socioeconomic status. Cochrane Database Syst Rev. 2025 Jan 27;1(1):CD015120. doi: 10.1002/14651858.CD015120.pub2. PMID 39868569
- [Derived] Notley C, Gentry S, Livingstone-Banks J, Bauld L, Perera R, Conde M, Hartmann-Boyce J. Incentives for smoking cessation. Cochrane Database Syst Rev. 2025 Jan 13;1(1):CD004307. doi: 10.1002/14651858.CD004307.pub7. PMID 39799985
- [Derived] Halpern SD, French B, Small DS, Saulsgiver K, Harhay MO, Audrain-McGovern J, Loewenstein G, Asch DA, Volpp KG. Heterogeneity in the Effects of Reward- and Deposit-based Financial Incentives on Smoking Cessation. Am J Respir Crit Care Med. 2016 Oct 15;194(8):981-988. doi: 10.1164/rccm.201601-0108OC. PMID 27064456
- [Derived] Halpern SD, French B, Small DS, Saulsgiver K, Harhay MO, Audrain-McGovern J, Loewenstein G, Brennan TA, Asch DA, Volpp KG. Randomized trial of four financial-incentive programs for smoking cessation. N Engl J Med. 2015 May 28;372(22):2108-17. doi: 10.1056/NEJMoa1414293. Epub 2015 May 13. PMID 25970009
- [Derived] French B, Small DS, Novak J, Saulsgiver KA, Harhay MO, Asch DA, Volpp KG, Halpern SD. Preference-adaptive randomization in comparative effectiveness studies. Trials. 2015 Mar 18;16:99. doi: 10.1186/s13063-015-0592-6. PMID 25887045